CLINICAL TRIAL: NCT04281342
Title: Prospective, Single-center, Randomized, Double-blind, Placebo- and Moxifloxacin-controlled, 4-way Crossover Phase 1 Study to Assess the Effect of Multiple Therapeutic and Supratherapeutic Doses of Aprocitentan on the QT Interval Duration in Healthy Subjects
Brief Title: To Study the Effect of Aprocitentan on the Electrical Activity of the Heart in Healthy Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-080-108; 2019-003617-34 (EudraCT Number)
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — aprocitentan

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized immediately prior to first study treatment administration on Day 1 Period 1 to one of 12 treatment sequences following a 3 × 4 × 4 Williams square design. Moxifloxacin will be open-label on Day 10 in one period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aprocitentan 25 mg (Experimental): Therapeutic dose level
  Interventions: Drug: Aprocitentan 25 mg
- Aprocitentan 100 mg (Experimental): Supratherapeutic dose level
  Interventions: Drug: Aprocitentan 100 mg
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo
- Moxifloxacin (Other)
  Interventions: Other: Moxifloxacin control to establish assay sensitivity

INTERVENTIONS:
Drug: Aprocitentan 25 mg — Repeated administration of a 25 mg oral dose of aprocitentan, once daily from Day 1 to Day 10, followed by 18 days of observation.
  Other Names: ACT-132577
  Arms: Aprocitentan 25 mg
Drug: Aprocitentan 100 mg — Repeated administration of a 100 mg oral dose of aprocitentan, once daily from Day 1 to Day 10, followed by 18 days of observation.
  Other Names: ACT-132577
  Arms: Aprocitentan 100 mg
Drug: Matching placebo — Repeated administration of an oral dose of aprocitentan-matching placebo, once daily from Day 1 to Day 10, followed by 18 days of observation.
  Arms: Matching placebo
Other: Moxifloxacin control to establish assay sensitivity — Repeated administration of an oral dose of aprocitentan-matching placebo, once daily from Day 1 to Day 9. On Day 10, oral administration of one single 400 mg moxifloxacin tablet open-label, followed by 18 days of observation.
  Arms: Moxifloxacin

SUMMARY:
To demonstrate that multiple-dose administration of oral therapeutic and supratherapeutic doses of aprocitentan do not have a clinically relevant effect on the QT interval.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Ability to communicate well with the investigator, in a language understandable to the subject, and to understand and comply with the requirements of the study.
* No clinically significant findings on the physical examination at screening.
* Body mass index 18.0 to 30.0 kg/m2 (inclusive) at screening.
* Systolic blood pressure 90-140 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 50-90 bpm (all inclusive), measured on the same arm, after 5 minutes in the supine position at screening.
* 12-lead safety ECG: QTcF less than 450 ms for male subjects and less than 470 ms for female subjects, QRS less than 110 ms, PR less than 220 ms, and resting HR greater than 50 bpm and less than 90 bpm with no clinically relevant abnormalities on 12-lead ECG after at least 5 min in the supine position at Screening and on Day 1 pre-dose of Period 1.
* No clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry) at screening.
* Negative results from urine drug screen, urine cotinine test, and breath alcohol tests at screening and on Day -1 of each period.
* A woman of childbearing potential (WoCBP) is eligible only if the following applies:

  * Negative serum pregnancy test at screening.
  * Negative urine pregnancy test on Day -1 of each period.
  * Agreement to consistently and correctly use a highly effective method of contraception from screening up to at least 30 days after last study treatment administration in the last period with in-between periods included.
* Women of non-childbearing potential (WoNCBP) must meet at least one of the following criteria:

  * Previous bilateral salpingectomy, salpingo-oophorectomy or hysterectomy,
  * Confirmed premature ovarian failure,
  * Post-menopausal.

Exclusion Criteria:

* Pregnant or lactating women.
* Previous exposure to aprocitentan or macitentan.
* Known hypersensitivity to aprocitentan or macitentan or any of the drug product excipients, or treatments of the same class.
* Any contraindication or known hypersensitivity to moxifloxacin or any of the drug product excipients or to other fluoroquinolone antibiotics.
* Known hypersensitivity or allergy to natural rubber latex.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation of the study.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 2 weeks or 5 t½ (whichever is longer) prior to first study treatment administration with the exception of contraceptives in female subjects.
* History or presence of rhythm disorders (e.g., sinoatrial heart block, sick-sinus syndrome, second- or third-degree atrioventricular block, long QT syndrome, symptomatic bradycardia, atrial flutter, or atrial fibrillation) or hypokalemia.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change from baseline in QT interval corrected with Fridericia's formula (ΔΔQTcF) | Multiple predefined time points related to study treatment administration on Day 1 and Day 10 to 11 of each treatment.

SECONDARY OUTCOMES:
Aprocitentan trough plasma concentrations (Ctrough) | Day 2 to Day 9
Aprocitentan plasma Cmax, first dose | Pre-defined times on the first dosing day (Day 1) up to 15 hours after last dose
Aprocitentan plasma Cmax, steady state | Pre-defined times on the last dosing day (Day 10) up to 15 hours after last dose
Area under the plasma concentration-time curve (AUCτ) during a dosage interval (τ) of aprocitentan | Day 1 to Day 10
Aprocitentan attainment of steady-state conditions | Day 1 to Day 10
Accumulation index between the first and the last dosing day of aprocitentan | Day 1; Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No